CLINICAL TRIAL: NCT00902694
Title: Randomized Trial Of Achieving Healthy Lifestyles In Psychiatric Rehabilitation
Brief Title: Randomized Trial Of Achieving Healthy Lifestyles In Psych Rehabilitation
Acronym: ACHIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH080964 (NIH); R01MH080964 (NIH); DAHBR 96-BHB; NIMH R01MH080964
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Results first posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Overweight and Obesity
Keywords: Serious Mental Illness; Weight Loss
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACHIEVE Intervention (Experimental): Group and individual weight counseling and group physical activity classes for 18 months.
  Interventions: Behavioral: ACHIEVE Intervention
- Control (Other): Control arm receives group health classes quarterly with topics not related to weight
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: ACHIEVE Intervention — Group and individual weight loss counseling and group physical activity classes for 18 months
  Arms: ACHIEVE Intervention
Other: Control — group health classes quarterly with topics not related to weight
  Arms: Control

SUMMARY:
This study will determine whether a behavioral weight loss intervention including dietary counseling and exercise is effective in helping people with serious mental illnesses lose weight.

DETAILED DESCRIPTION:
The objective of this study is to perform a randomized clinical trial (ACHIEVE) to definitively test the efficacy of an innovative, practical intervention to accomplish weight loss in overweight and obese persons with SMI. This multi-site trial will enroll consumers with SMI who attend ten psychiatric rehabilitation centers in Maryland and randomize participants to the ACHIEVE intervention or control. Intervention participants will receive group and individual weight loss counseling sessions and group physical activity classes. Co-primary outcomes will be change in weight from baseline to 6 and 18 months.

ELIGIBILITY:
Age 18 and older;

* Overweight, defined by Body Mass Index at least 25.0 kg/m2;
* Able and willing to give informed consent and participate in the intervention;
* On the same psychiatric medications within the 30 days before baseline weight (dose changes allowed;)
* Able to attend at least 2 intervention sessions per week during initial 6-month phase;

Exclusion criteria

* Contraindication to weight loss

  * Receiving active cancer treatment (radiation/chemotherapy)
  * Liver failure
  * History of anorexia nervosa;
* Cardiovascular event (unstable angina, myocardial infarction) within previous 6 months;
* Prior or planned bariatric surgery;

Use of prescription weight loss medication or over-the-counter orlistat within 3 months

if participant does not agree to stop taking it;

* Twenty pound or greater weight loss in 3 months prior to baseline, as documented by staff measurement;
* Inability to walk to participate in exercise class;
* Pregnant or planning a pregnancy during study period. Nursing mothers would need approval from physician;
* Alcohol or substance use disorder either: 1) active and determined to be incompatible with participation in the intervention through discussion with program staff; or 2) new abstinence from alcohol or substance use disorder in past 30 days;
* Planning to leave rehabilitation center within 6 months or move out of geographic area within 18 months;
* Investigator judgment (e.g., for concerns over safety, adherence or follow-up);
* Weight greater than 400 pounds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2008-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail L. Daumit, MD, MHS, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Prohealth, Baltimore, Maryland, United States

REFERENCES:
- [Background] Casagrande SS, Jerome GJ, Dalcin AT, Dickerson FB, Anderson CA, Appel LJ, Charleston J, Crum RM, Young DR, Guallar E, Frick KD, Goldberg RW, Oefinger M, Finkelstein J, Gennusa JV 3rd, Fred-Omojole O, Campbell LM, Wang NY, Daumit GL. Randomized trial of achieving healthy lifestyles in psychiatric rehabilitation: the ACHIEVE trial. BMC Psychiatry. 2010 Dec 13;10:108. doi: 10.1186/1471-244X-10-108. PMID 21144025
- [Derived] Janssen EM, Jerome GJ, Dalcin AT, Gennusa JV 3rd, Goldsholl S, Frick KD, Wang NY, Appel LJ, Daumit GL. A cost analysis of implementing a behavioral weight loss intervention in community mental health settings: Results from the ACHIEVE trial. Obesity (Silver Spring). 2017 Jun;25(6):1006-1013. doi: 10.1002/oby.21836. Epub 2017 Apr 11. PMID 28398006
- [Derived] Daumit GL, Dickerson FB, Wang NY, Dalcin A, Jerome GJ, Anderson CA, Young DR, Frick KD, Yu A, Gennusa JV 3rd, Oefinger M, Crum RM, Charleston J, Casagrande SS, Guallar E, Goldberg RW, Campbell LM, Appel LJ. A behavioral weight-loss intervention in persons with serious mental illness. N Engl J Med. 2013 Apr 25;368(17):1594-602. doi: 10.1056/NEJMoa1214530. Epub 2013 Mar 21. PMID 23517118

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACHIEVE Intervention | Control
Started | 144 | 147
Completed | 137 | 142
Not Completed | 7 | 5
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Censored per protocol | 3 | 1
Not completed — Pregnancy | 1 | 1
Not completed — Incarceration | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ACHIEVE Intervention | Control | Total
Number analyzed (Participants) | 144 | 147 | 291
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 137 | 145 | 282
  >=65 years | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (11.5) | 44.1 (11.0) | 45.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 72 | 146
  Male | 70 | 75 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 13
  Not Hispanic or Latino | 139 | 139 | 278
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 52 | 59 | 111
  White | 82 | 81 | 163
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 144 | 147 | 291
primary psychiatric diagnosis [Count of Participants; unit: Participants]
  schizophrenia | 44 | 41 | 85
  schizoaffective disorder | 41 | 43 | 84
  bipolar disorder | 28 | 36 | 64
  major depressive disorder | 18 | 17 | 35
  other | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight Loss in Kilograms (kg)
Description: Change is from baseline to 6 months and baseline to 18 months
Time Frame: 6 and 18 months
Measure: Mean (95% Confidence Interval); unit: kg
Arm/Group | ACHIEVE Intervention | Control
Number analyzed (Participants) | 144 | 147
kg
  baseline to 6 month change | -1.8 [-2.5 to -1.0] | -0.3 [-1.0 to 0.5]
  baseline to 18 month change | -3.4 [-4.7 to -2.1] | -0.2 [-1.7 to 1.3]
Statistical Analysis 1: Comparison: ACHIEVE Intervention vs Control; 6 month intervention versus control; Test type: Superiority; Mean Difference (Net) = -1.5, 95% CI 2-sided [-2.6 to -0.4]
Statistical Analysis 2: Comparison: ACHIEVE Intervention vs Control; 18 month intervention versus control; Test type: Superiority; Mean Difference (Net) = -3.2, 95% CI 2-sided [-5.1 to -1.2]

2. Secondary Outcome: Minutes Cycled During Cycle Ergometry Testing
Description: Minutes cycled during standardized cycle ergometry testing protocol; higher number of minutes cycled indicates better outcome.
Time Frame: Baseline, 6 and 18 months
Population: Cycle ergometry test was not completed for those who completed data collection off-site where no bicycle ergometer was available. Results are not modeled.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | ACHIEVE Intervention | Control
Number analyzed (Participants) | 136 | 142
minutes
  baseline | 6.95 (2.64) | 6.86 (2.86)
  6 month | 7.12 (2.86) | 6.91 (2.82)
  18 month | 7.19 (3.03) | 6.79 (2.60)

3. Secondary Outcome: Change in Waist Circumference in Centimeters (cm)
Description: Change in waist circumference in centimeters (cm) from baseline to 18 months
Time Frame: Measured at baseline, 6 and 18 months
Population: Reported for those who completed this measure at these follow-up data points.
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | ACHIEVE Intervention | Control
Number analyzed (Participants) | 113 | 124
cm
  baseline to 6 month change | -1.5 [-2.6 to -0.4] | 0.5 [-0.7 to 1.7]
  baseline to 18 month change | -2.2 [-3.8 to -0.7] | -1.9 [-4.1 to 0.3]
Statistical Analysis 1: Comparison: ACHIEVE Intervention vs Control; 6 month intervention versus control; Test type: Superiority; Mean Difference (Net) = -2.0, 95% CI 2-sided [-3.6 to -0.4]
Statistical Analysis 2: Comparison: ACHIEVE Intervention vs Control; 18 month intervention versus control; Test type: Superiority; Mean Difference (Net) = -1.9, 95% CI 2-sided [-4.1 to 0.3]

4. Secondary Outcome: Change in Systolic and Diastolic Blood Pressure (mmHg)
Description: Change in systolic and diastolic blood pressure (mmHg) from baseline to 18 months
Time Frame: Measured at baseline, 6 and 18 months
Population: Reported for those who completed this measure at these follow-up data points.
Measure: Mean (95% Confidence Interval); unit: mmhg
Arm/Group | ACHIEVE Intervention | Control
Number analyzed (Participants) | 134 | 140
mmhg
  baseline to 6 month systolic change | -2.5 [-4.7 to -0.2] | -2.1 [-3.8 to -0.4]
  baseline to 6 month diastolic change | -0.7 [-2.0 to 0.7] | -0.9 [-2.2 to 0.3]
  baseline to 18 month systolic change | -1.1 [-3.5 to 1.3] | -2.7 [-4.8 to -0.7]
  baseline to 18 month diastolic change | -0.6 [-2.2 to 0.9] | -1.9 [-3.3 to -0.4]
Statistical Analysis 1: Comparison: ACHIEVE Intervention vs Control; 6 month systolic intervention versus control; Test type: Superiority; Mean Difference (Net) = -0.4, 95% CI 2-sided [-3.2 to 2.4]
Statistical Analysis 2: Comparison: ACHIEVE Intervention vs Control; 6 month diastolic intervention versus control; Test type: Superiority; Mean Difference (Net) = 0.2, 95% CI 2-sided [-1.6 to 2.1]
Statistical Analysis 3: Comparison: ACHIEVE Intervention vs Control; 18 month systolic intervention versus control; Test type: Superiority; Mean Difference (Net) = 1.6, 95% CI 2-sided [-1.6 to 4.8]
Statistical Analysis 4: Comparison: ACHIEVE Intervention vs Control; 18 month diastolic intervention versus control; Test type: Superiority; Mean Difference (Net) = 1.2, 95% CI 2-sided [-0.9 to 3.4]

5. Secondary Outcome: Change in Lipids (Total Cholesterol, LDL, HDL and Triglyceride (mg/dL)
Description: Change in Lipids (total cholesterol, LDL, HDL and Triglyceride (mg/dL) from baseline to 18 months
Time Frame: Measured at baseline, 6 and 18 months
Population: Reported for those who completed this measure at these follow-up data points.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | ACHIEVE Intervention | Control
Number analyzed (Participants) | 124 | 125
mg/dl
  baseline to 6 month total chol change | -4.8 [-9.8 to 0.2] | -1.9 [-6.8 to 3.0]
  baseline to 18 month total chol change | -5.6 [-11.8 to 0.6] | -0.3 [-7.8 to 7.1]
  baseline to 6 month LDL chol change | -3.8 [-8.0 to 0.5] | -2.5 [-7.2 to 2.1]
  baseline to 18 month LDL chol change | -5.5 [-10.7 to -0.2] | -0.9 [-7.6 to 5.8]
  baseline to 6 month HDL chol change | 0.2 [-1.0 to 1.4] | 0.8 [-1.2 to 2.8]
  baseline to 18 month HDL chol change | 0.6 [-1.2 to 2.3] | -0.1 [-1.8 to 1.7]
  baseline to 6 month TRIG change | -6.3 [-16.6 to 3.9] | -0.8 [-15.6 to 14.0]
  baseline to 18 month TRIG change | 3.5 [-15.1 to 22.1] | 5.0 [-12.4 to 22.4]
Statistical Analysis 1: Comparison: ACHIEVE Intervention vs Control; 6 month total chol intervention versus control; Test type: Superiority; Mean Difference (Net) = -2.9, 95% CI 2-sided [-9.9 to 4.1]
Statistical Analysis 2: Comparison: ACHIEVE Intervention vs Control; 18 month total chol intervention versus control; Test type: Superiority; Mean Difference (Net) = -5.2, 95% CI 2-sided [-14.9 to 4.4]
Statistical Analysis 3: Comparison: ACHIEVE Intervention vs Control; 6 month LDL chol intervention versus control; Test type: Superiority; Mean Difference (Net) = -1.2, 95% CI 2-sided [-7.5 to 5.1]
Statistical Analysis 4: Comparison: ACHIEVE Intervention vs Control; 18 month LDL chol intervention versus control; Test type: Superiority; Mean Difference (Net) = -4.6, 95% CI 2-sided [-13.1 to 3.9]
Statistical Analysis 5: Comparison: ACHIEVE Intervention vs Control; 6 month HDL chol intervention versus control; Test type: Superiority; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.9 to 1.7]
Statistical Analysis 6: Comparison: ACHIEVE Intervention vs Control; 18 month HDL intervention versus control; Test type: Superiority; Mean Difference (Net) = 0.6, 95% CI 2-sided [-1.8 to 3.1]
Statistical Analysis 7: Comparison: ACHIEVE Intervention vs Control; 6 month TRIG intervention versus control; Test type: Superiority; Mean Difference (Net) = -5.5, 95% CI 2-sided [-23.5 to 12.4]
Statistical Analysis 8: Comparison: ACHIEVE Intervention vs Control; 18 month TRIG intervention versus control; Test type: Superiority; Mean Difference (Net) = -1.5, 95% CI 2-sided [-27.0 to 23.9]

6. Secondary Outcome: Framingham Cardiovascular Risk Score
Description: Higher score indicates greater cardiovascular risk. The score can range from 0-38 with higher scores yielding increased 10-year probability of stroke
Time Frame: Measured at baseline, 6 and 18 months
Population: Only included data for those participants who had all variables in calculation equation. Not modeled
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACHIEVE Intervention | Control
Number analyzed (Participants) | 143 | 146
score on a scale
  Baseline | 0.0999 (0.1027) | 0.0989 (0.0924)
  6 month | 0.1029 (0.1093) | 0.0991 (0.0953)
  18 month | 0.1035 (0.0972) | 0.0978 (0.0925)

7. Secondary Outcome: Health Status as Measured by the SF-12
Description: Health status reported for the SF-12 in two subscales-physical component summary (PCS) and the mental component summary (MCS). Subscale score ranges from 0-100 with higher scores indicating better physical or mental health.
Time Frame: Baseline, 6 and 18 months
Population: Reported for those who completed this measure at these follow-up data points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACHIEVE Intervention | Control
Number analyzed (Participants) | 144 | 147
score on a scale
  Baseline PCS score | 45.1 (10.6) | 43.4 (9.7)
  6 months PCS Score | 45.5 (10.4) | 43.8 (10.8)
  18 months PCS score | 46.2 (11.6) | 44.4 (10.1)
  Baseline MCS score | 45.0 (11.4) | 45.8 (10.2)
  6 months MCS score | 46.2 (10.8) | 44.4 (10.9)
  18 months MCS score | 45.1 (11.5) | 45.5 (11.2)

8. Secondary Outcome: Depression Assessed by Center for Epidemiologic Studies Depression Scale (CES-D)
Description: Total score range between 0 and 60, higher scores indicating more depressive symptoms
Time Frame: Baseline, 6 and 18 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ACHIEVE Intervention | Control
Number analyzed (Participants) | 144 | 147
score on a scale
  Baseline | 19.7 (11.3) | 20.1 (11.2)
  6 months | 18.7 (11.6) | 20.9 (11.5)
  18 months | 18.7 (11.0) | 19.5 (11.2)

ADVERSE EVENTS:
Time Frame: baseline through 18 months
Arm/Group | ACHIEVE Intervention | Control
All-Cause Mortality (participants affected / at risk) | 2/144 | 3/147
Serious Adverse Events (participants affected / at risk) | 42/144 | 47/147
Other Adverse Events (participants affected / at risk) | 0/144 | 0/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ACHIEVE Intervention (N=144) | Control (N=147)
psychiatric hospitalization (Psychiatric disorders) | 21 (31) | 30 (51)
medical hospitalizations (General disorders) | 26 (33) | 19 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No